CLINICAL TRIAL: NCT05274217
Title: Discovering Our Story, to Develop the Journey of Transformation
Brief Title: Journey of Transformation Curriculum for Native American Adolescents
Acronym: JOT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Significant revision of protocol inspired by site staff changes and site COVID delays
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Teresa Evans-Campbell, Associate Professor: School of Social Work, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00012676; 1R01DA050521-01A1 (NIH)
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Alcohol Use; Tobacco Use; Substance Use; Sexual Health
Keywords: Native American; American Indian; Adolescents
MeSH Terms: conditions — Alcohol Drinking; Tobacco Use; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: A randomized waitlist stepped wedge design with study participants recruited in staggered cohorts, with those in each annual recruitment wave receiving individual-level random assignment to either immediate intervention or waitlist control.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate group (Experimental): Study participants in the immediate group will be randomly assigned to start the intervention immediately at the beginning of the fall trimester.
  Interventions: Behavioral: Journey of Transformation-Native Youth Health Leadership Program curriculum
- Waitlist group (Experimental): Study participants in the waitlist group will be randomly assigned to start the intervention at the beginning of the winter trimester.
  Interventions: Behavioral: Journey of Transformation-Native Youth Health Leadership Program curriculum

INTERVENTIONS:
Behavioral: Journey of Transformation-Native Youth Health Leadership Program curriculum — Curriculum activities will include traditional storytelling and other Native American cultural arts activities (i.e., drum making, film making), as well as Traditional Ecological Knowledge (TEK) activities and field trips. Curriculum content explains leadership skills and promotes healthy decision-making around substance use and sexual health.

SUMMARY:
The investigators will conduct a waitlist control trial to test the efficacy of the Journey of Transformation-Native Youth Health Leadership Program (JOT) in terms of delaying or reducing tobacco and other substance use and improving sexual health.

DETAILED DESCRIPTION:
This study assesses a new curriculum that will be available to students in the ninth grade. The lessons will include traditional storytelling and other Native American cultural arts activities (i.e., drum making, film making, field trips), as well as Traditional Ecological Knowledge (TEK) activities. This study also assesses how well the curriculum explains leadership skills, Native American cultural arts, the natural environment, and promotes healthy decision-making around health and relationships.

Participants are randomly assigned to a health class that starts the curriculum in the fall or to a health class that will start the curriculum in the winter. Participants will:

Week 1. Take a 30-40 minute online survey about healthy relationships, drug use, youth leadership skills and connecting with Native communities.

Weeks 1-3. Meet with a counselor up to two times to set goals around health, healthy relationships and how to reduce or avoid alcohol, tobacco, or other drug use.

Weeks 1 - 8 (months 1-2). As part of the health class, attend about 16 health sessions on healthy behaviors and health promotion. Learn new skills around youth leadership, storytelling, and traditional health practices. The sessions will highlight connecting to tribal traditions.

Month 3. Take an online check-in survey via a link sent to participants' email address.

Month 6. Take an online check-in survey via a link sent to participants' email address.

Month 12. Take an online check-in survey via a link sent to participants' email address.

Optional after school activities Week 9-16 (months 3-4). Attend a once-a-month activity to help build leadership skills. Activities are between 1-2 hours after school and include drum making, film making, creating a storytelling vest that incorporates cultural symbols, and up to two outdoor field trips. The field trips are to places of cultural significance near the school and involve a 30-45 minute hike.

Week 16 (month 4). Meet with the study counselor for a session to revise goals for health and community leadership.

Week 9-24 (months 3 - 6). Attend a 2-hour digital storytelling training and three-monthly planning sessions to prepare for an optional digital storytelling leadership night. The story can be about what has been learned about health promotion, traditional health practices, and to celebrate participants' health leadership journey.

Week 25 (month 6). Attend the leadership night and present digital stories.

ELIGIBILITY:
Inclusion Criteria:

* Between 13 years of age and 16 years of age
* Attending an off-reservation boarding school in the ninth grade at time of enrollment

Exclusion Criteria:

* Under 13 years old, or over 16 years old
* Does not attend an off-reservation boarding school in the ninth grade at time of enrollment

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa A Evans-Campbell, MSW, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified individual participant data (IPD) will be available after Institutional Review Board (IRB) and agency approval.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: De-identified data will be available for 12 months after publication of the main findings manuscript. Other resources, such as training materials and the curriculum, will be available after demonstration of their efficacy.
Access Criteria: Contact PI for access.

REFERENCES:
- [Background] National Institute on Drug Abuse, University of Michigan, Institute for Social Research. (2016). Monitoring the Future, 2016 (Combined Forms - Part B). Ann Arbor, MI: Institute for Social Research, University of Michigan.
- [Background] Hansen WB, Paskett ED, Carter LJ. The Adolescent Sexual Activity Index (ASAI): a standardized strategy for measuring interpersonal heterosexual behaviors among youth. Health Educ Res. 1999 Aug;14(4):485-90. doi: 10.1093/her/14.4.485. PMID 10557519
- [Background] Miech, Richard A., Johnston, Lloyd D., Bachman, Jerald G., O'Malley, Patrick M., Schulenberg, John E., and Patrick, Megan E. Monitoring the Future: A Continuing Study of American Youth (8th- and 10th-Grade Surveys), 2020. Inter-university Consortium for Political and Social Research [distributor], 2021-10-26. https://doi.org/10.3886/ICPSR38189.v1
- [Background] Belgrave FZ, Reed MC, Plybon LE, Corneille M. The impact of a culturally enhanced drug prevention program on drug and alcohol refusal efficacy among urban African American girls. J Drug Educ. 2004;34(3):267-79. doi: 10.2190/H40Y-D098-GCFA-EL74. PMID 15648887
- [Background] Petosa R, Jackson K. Using the health belief model to predict safer sex intentions among adolescents. Health Educ Q. 1991 Winter;18(4):463-76. doi: 10.1177/109019819101800405. PMID 1757268

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Group | Waitlist Group
Started | 33 | 0
Completed | 22 | 0
Not Completed | 11 | 0
Not completed — Study terminated. | 11 | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated due to a significant revision of protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Group | Waitlist Group | Total
Number analyzed (Participants) | 22 | 0 | 22
Age, Continuous [Mean (Full Range); unit: years] | 14.4 [13.0 to 16.0] |  | 14.4 [13.0 to 16.0]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 13 |  | 13
  Sex: Male | 8 |  | 8
  Sex: Unknown | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 22 |  | 22
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 0 |  | 0
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 |  | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Patterns of 30 Day Substance Use Assessed by Self-report
Description: Patterns of substance use (Monitoring the Future [MTF] 30-day self-report assessed on an ordinal scale [0 occasions, 1-2 occasions, 3-5 occasions, 6-9 occasions, 10-19 occasions, 20-39 occasions, 40 or more occasions]). Substances include tobacco, alcohol, marijuana, stimulants, inhalants, opioids, and other drugs.
Time Frame: Baseline to 3-month (post-intervention) follow-up; Baseline to 6-month follow-up; Baseline to 12-month follow-up (immediate group only)
Population: Outcome data is not available due to study termination at baseline. Therefore, post-intervention and follow-up data were not collected.
Arm/Group | Immediate Group | Waitlist Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Sexual Behavior Assessed by the Adolescent Sexual Activity Index (ASAI)
Description: The Adolescent Sexual Activity Index (ASAI) is a 13-item index which assesses pre-coitus sexual behaviors and produces an 11-point scale from 0-10 (Hansen et al., 1999).
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Immediate Group | Waitlist Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Intentions to Use Alcohol, Cigarettes, and Marijuana in the Next Year (Assessed by Monitoring the Future [MTF])
Description: Assess intention to use alcohol, cigarettes, and marijuana in the next year (3 items) on a 5-point scale (I have already tried [substance], I definitely will, I probably will, I probably will not, I definitely will not). Scores are summed and standardized on a scale of 0 to 100 percent.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Immediate Group | Waitlist Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in the Specific Event Drug and Alcohol Refusal Self-Efficacy (SEDARE) Measure
Description: The Specific Event Drug and Alcohol Refusal Self-Efficacy (SEDARE) measure captures the perceived likelihood that youth will use drugs and alcohol in specific situations on a 3-point scale (Yes, No, Unsure). Higher scores reflect higher perceived ability to refuse alcohol or drugs.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Immediate Group | Waitlist Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in the Health Belief Model-Intentions for Safer Sex Intentions (HBMI) (Lux & Petosa, 1994)
Description: 7 items will be used to predict safer sex intentions on a 5-point Likert scale (strongly agree to strongly disagree, where 1 is strongly agree).
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Immediate Group | Waitlist Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Description: We used the clinicaltrials.gov definitions of "adverse event" and "serious adverse event."
Arm/Group | Immediate Group | Waitlist Group
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/0
Other Adverse Events (participants affected / at risk) | 0/33 | 0/0

LIMITATIONS AND CAVEATS:
Early termination of trial led to no post outcomes. No subjects were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT05274217/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT05274217/SAP_001.pdf
  • Informed Consent Form: Assent Form (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT05274217/ICF_002.pdf
  • Informed Consent Form: Parent / Guardian Permission Form (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT05274217/ICF_003.pdf